CLINICAL TRIAL: NCT02946437
Title: Short Term Application of Sevoflurane in Patients With Subarachnoid Haemorrhage: a Feasibility and Safety Study
Brief Title: Sevoflurane in Subarachnoidal Haemorrhage
Acronym: Sevoflurane
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Patients failed to be enrolled because of tight exclusion criteria.
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Emanuela Keller, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0397; 2015DR2134 (Other: Swissmedic)
Record Dates: First submitted 2016-10-07; First posted 2016-10-27 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Subarachnoid Haemorrhage (SAH)
Keywords: severe SAH; prevention of vasospasm and/ or brain oedema; Sevoflurane; Postconditioning
MeSH Terms: conditions — Subarachnoid Hemorrhage; Brain Edema | interventions — Sevoflurane; Propofol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sevoflurane (Experimental): Sevoflurane postconditioning will start after the bleeding source is excluded by coiling or clipping as soon as the patient returns to the ICU and will be continued for 4 hours. 0.5-1.5vol% sevoflurane will be administrated into the ventilation circuit by a MIRUS™System.
  The used dose (0.5-1.5vol%) is a lower dose as used for anaesthesia for a surgical intervention (0.5-3vol%), but high enough to provide sufficient sedation.
  Interventions: Drug: Sevoflurane; Device: MIRUS™System
- Propofol or Midazolam (Active Comparator): Propofol or midazolam will be administrated intravenously before and after the postconditioning with sevoflurane as in the standard sedation regimen of the Neurointensive Care Unit, University Hospital Zurich (propofol 0.3-4.0mg/kg/h cont. i.v.; midazolam 0.03-0.2mg/kg/h cont. i.v.)
  Interventions: Drug: Propofol; Drug: Midazolam
- MIRUS™System (Other): MIRUS™ is a newly developed device, considered as vaporizer system, which can be used in the setting of operating rooms or in intensive care units. The MIRUS™System is successfully in use in daily clinical practice. This type of device is similar to the well-known AnaConDa® system (AnaConDa®, Sedana Medical, Uppsala, S) with several advantages. Since 2005 the anaesthetic-conserving device AnaConDa® facilitates, from a technical viewpoint, the routine use of volatile anaesthetics in intensive care patients as part of prolonged sedation, using ICU ventilators (Soukup J et al., 2009). The MIRUS™System forms a closed loop. It measures the end-tidal concentration of the anaesthetic gas and governs the application of the anaesthetic gas according to these values and the ventilation parameters.
  Interventions: Drug: Sevoflurane; Device: MIRUS™System

INTERVENTIONS:
Drug: Sevoflurane — Postconditioning with sevoflurane (0.5-1.5vol%) for 4 hours after coiling or clipping of cerebral aneurysm in patients with severe SAH
  Other Names: Sevorane®
  Arms: MIRUS™System; Sevoflurane
Drug: Propofol — Before and after postconditioning with sevoflurane the patients will be sedated with intravenous sedatives (midazolam or propofol). The quality of sedation before the postconditioning (propofol or midazolam) will be compared to the sedation one hour after starting the postconditioning (sevoflurane) in the same patient.
  Other Names: Disoprivan®
  Arms: Propofol or Midazolam
Drug: Midazolam — Before and after postconditioning with sevoflurane the patients will be sedated with intravenous sedatives (midazolam or propofol). The quality of sedation before the postconditioning (propofol or midazolam) will be compared to the sedation one hour after starting the postconditioning (sevoflurane) in the same patient.
  Other Names: Dormicum®
  Arms: Propofol or Midazolam
Device: MIRUS™System — The MIRUS™System is the normally used standard equipment for the administration of volatile anaesthetics to patients.
  Arms: MIRUS™System; Sevoflurane

SUMMARY:
Feasibility and safety of short term application of sevoflurane in patients with SAH treated with aneurysm coiling or clipping in the setting of a neurointensive care unit.

DETAILED DESCRIPTION:
After admission to the ICU, before the coiling / clipping intervention has been performed, the patients are screened for eligibility. When the patients are coming back to the ICU, after successful aneurysm coiling or clipping, data of artificial ventilation, systemic and other cerebral parameters will be collected continuously by online monitoring, starting at baseline and stopping at discharge of the ICU. Sevoflurane will be vaporized and administrated by the MIRUS™System directly to the inspiratory part of the ventilation circuit for the next 4 hours. In the following 14 days of the stay on the ICU, standard monitoring parameters, the appearance of vasospasm and brain oedema will be recorded. Besides the continuous online monitoring, laboratory assessment will be performed daily. At day 7±2 and day 14±2 after bleeding a MRI or CT examination will be performed, according to the clinical condition of the patient, to detect secondary brain injuries, as ischemia or brain oedema. At ICU discharge, the neurological outcome will be assesses applying GOS.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 18-85 years
* Patients with severe aneurysmal SAH, Hunt/Hess 3 to 5.
* The ruptured aneurysm is successfully excluded with coiling or clipping
* Sedation and mechanical ventilation necessary due to the clinical situation
* ICP monitoring in use due to the clinical situation
* ICP < 20mmHg without medical treatment
* Systolic blood pressure values (BP syst) > 120 mmHg with no need for catecholamines
* Female patients of childbearing potential with negative pre-treatment serum pregnancy test
* Informed consent obtained

Exclusion Criteria:

* Significant kidney disease, defined as plasma creatinine >120 µmol/l
* Significant liver disease, defined as Aspartate-Aminotransferase (AST) >200 U/l
* Significant elongation of the QTc interval: female < 470 msec/ male < 450 msec; based on 'Bazett's Formula'
* History of epilepsia and/ or occurring seizures with aneurysm rupture
* Pneumocephalus after surgery excluded by CT scan performed immediately after clipping
* History of allergic disorders
* History for, or relatives with a history for malignant hyperthermia
* History or signs for neuromuscular disease
* Pre-existing disability
* Patients participating in an interventional clinical trial within the last 30 days before start of treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility: Incidence of concerns/problems in the use of sevoflurane by intensivist and ICU nurse at the stopping of sevoflurane postconditioning. | 4 hours
  * Incidence of concerns of users in relation to the application of standard sedation with propofol or midazolam
  * Incidence of complications with sevoflurane preparation, sevoflurane application, MIRUS™-installation, MIRUS™-function, MIRUS™-removal
  * User friendliness compared to settings for artificial ventilation supplemented with NO

SECONDARY OUTCOMES:
Quality of sedation | 5 hours
  * Incidence of insufficient sedation during postconditioning with sevoflurane, measured with:
    * Ramsay Sedation Scale (RSS <2)
    * Richmond Agitation-Sedation Scale (RASS >0)
    * Bispectral index (BIS >30)
    * Incidence of use of additional sedative medication as midazolam, propofol
  * in relation to the sedation regimen before and after the postconditioning (dose and use of additional sedative medication as midazolam, propofol)
Neuroprotective effects | 14 days
  * Number of days during the 14 days monitoring period with signs of DIND
    * incidence of new neurological deficits on daily clinical visits
    * incidence of 2 consecutive metabolic crisis identified by microdialysis, defined as lactate/pyrovate-ratio (L/P-ratio) >40
    * incidence of PtiO2 <20mmHg at least 60 minutes- immediately before the measurement
    * incidence of new perfusion deficits in perfusion-CT and/ or -MRI, new infarctions in contrast enhanced CT/ MRI
  * Neurological outcome (GOS) will be assessed at ICU discharge and compared to data from the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Keller, MD Prof., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No